CLINICAL TRIAL: NCT04037917
Title: The CorNeat EverPatch - a First-In-Man Clinical Study for Demonstrating the Safety of a Synthetic Tissue Substitute for Concealment of Artificial Implants and Glaucoma Tube Shunts
Brief Title: First-In-Man Study for an Ophthalmic Synthetic Tissue Substitute
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: CorNeat Vision Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-001
Record Dates: First submitted 2019-05-15; First posted 2019-07-30 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2022-04

CONDITIONS: Glaucoma Eye; Tissue Breakdown

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Synthetic Tissue Substitute (Experimental): Corneat EverPatch - Synthetic Tissue Substitute for Covering Ophthalmic Implants
  Interventions: Device: CorNeat EverPatch

INTERVENTIONS:
Device: CorNeat EverPatch — Covering Ophthalmic Implants

SUMMARY:
Study Name: The CorNeat EverPatch - a First-In-Man Clinical Study for demonstrating the Safety of a Synthetic Tissue Substitute for concealment of artificial implants and glaucoma tube shunts

Objective: The objective of this clinical trial is to demonstrate the Safety of the Corneat Everpatch for concealment of artificial implants and glaucoma tube shunts

The study will consist 10 subjects requiring concealment of a glaucoma shunt or other ophthalmic implant. Eligible subjects who signs an ICF will be enrolled to the study. Subjects will be implanted with the Corneart EverPatch as part of a glaucoma shunt surgery or during a corrective surgery to repair a breached conjunctiva over an implanted device. Subjects will be monitored for a period of 12 months post-op during which follow up visits will occur at 1 week, 1, 2, 3, 6, 9 & 12 months following surgery including clinical examination of the operated eye using slit-lamp biomicroscopy and imaging using OCT or UBM (will be performed only at the 6 & 12 months follow up visits).

DETAILED DESCRIPTION:
Study Name: The CorNeat EverPatch - a First-In-Man Clinical Study for demonstrating the Safety of a Synthetic Tissue Substitute for concealment of artificial implants and glaucoma tube shunts

Objective: The objective of this clinical trial is to demonstrate the Safety of the Corneat Everpatch for concealment of artificial implants and glaucoma tube shunts

Study endpoints:

Primary Safety Endpoint:

The frequency of all Unanticipated Adverse Device-related Events (UADE) or treatment-related adverse events, during and following implantation and follow-up for up to 12 months will be 10% or less.

Effectiveness Endpoints:

Primary: Conjunctival integrity at the implantation site will be 90% or more. Secondary: Stability in patch dimensions, less than 10% change (length, projected width and thickness) measured by OCT after 1-week and follow-up for up to 12 months post-implantation in 90% of the implanted patients.

Intended uses: The CorNeat EverPatch intended use is concealment of artificial ophthalmic implants and glaucoma tube shunts.

The clinical investigation of the CorNeat EverPatch device is essential to validate its safety and efficacy in its target implantation site and to substantiate regulatory clearance. Clinical investigation of a medical device must be in compliance with Good Clinical Practice as set forth in ISO 14155, which addresses good clinical practices for the design, conduct, recording and reporting of clinical investigations carried out in human subjects for the purpose of assessing the safety and performance of medical devices for regulatory purposes, as well as applicable local laws and regulations.

Study Population: 10 subjects requiring concealment of artificial ophthalmic implants and glaucoma tube shunts. Unilateral and bi-lateral. The device can be implanted in patients' right or left eye (selection according to Principle Investigator's discretion).

Study Duration: Subjects will be followed-up for 12 months from device implantation date.

Visit Schedule:

• Screening: Day 0-7, Subjects will sign an Informed Consent Form (ICF) on screening visit and baseline assessments for clinical condition, concomitant medication and medical history data will be performed.

• Implantation: Implantation day will be recorded as day 0; enrollment day.

• Follow up visits at 1 week, 1, 2, 3, 6, 9 & 12-month post-op (total of 7 follow up visits).

At each follow up visit, subjects will be evaluated for: (i) conjunctival integrity; (ii) device dimensions, (iii) clinical evaluation; (iv) device retention and (v) any clinically necessary interim safety exam per PI decision. Additionally, at 6 & 12 months post-op, subjects will undergo an imaging evaluation of the device's dimensions (either by UBM or OCT).

Safety Assessment: A record of UADE as well as incidence and nature of Serious Adverse Events (SAE) will be recorded. Incidence and nature of Adverse Events (AE) will be collected throughout the study starting from implantation. The following types of events are outside of this category:

(i) Adverse events related to the disease such as glaucoma and not caused by implant concealment (ii) Adverse events related to the primary implant such as tube shunt blockage not related to implant concealment

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Aged ≥ 18 and ≤ 80 years on screening day
3. Concealment of an artificial ophthalmic implant or a glaucoma tube shunt is indicated.
4. Candidates must have the ability and willingness to attend all scheduled visits and comply with all study procedures
5. Adequate tear film and lid function
6. Visual acuity of light perception or better
7. Female patients of childbearing age must agree to use a method of contraception and have negative pregnancy test at screening. An effective method of contraception must be used throughout the study.

Exclusion Criteria:

1. Current retinal detachment
2. Active ocular or orbital infection
3. History or evidence of severe inflammatory eye diseases (i.e. uveitis, retinitis, scleritis) in one or both eyes within 6 months prior to planned implantation
4. History of ocular or periocular malignancy
5. History of extensive keloid formation
6. Any known intolerance or hypersensitivity to topical anesthetics, mydriatics, or component of the device
7. Signs of current infection, including fever and current treatment with antibiotics
8. Severe generalized disease that results in a life expectancy shorter than a year
9. Any clinical evidence that the investigator feels would place the subject at increased risk with the placement of the device
10. Currently pregnant or breastfeeding
11. Participation in any study involving an investigational drug or device within the past 30 days or 5 half-lives of the drug (whichever longer) or ongoing participation in a study with an investigational drug or device
12. Intraoperative complication that would preclude implantation of the study device.
13. Any traumatic perforation
14. Tissue gaps/weaknesses, resulting either from traumatic, disease-related or iatrogenic damage
15. Loss of scleral integrity where use of tissue or substitutes is indicated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Number of treatment-related adverse events | up to 12 months
  The frequency of all Unanticipated Adverse Device-related Events (UADE) or treatment-related adverse events

SECONDARY OUTCOMES:
Conjunctival integrity | up to 12 months
  Conjunctival integrity at the implantation should be 90% or more as measured by Slit lamp examination
Stability in patch dimensions | up to 12 months
  Stability in patch dimensions should show less than 10% change (length, projected width and thickness) measured by OCT after 1-week and follow-up for up to 12 months post-implantation in 90% of the implanted patients

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (2):
  - Prism Eye Institute, Oakville, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
- Hospital Foundation Adolphe De Rothschild, Paris, France
- Kenya (3):
  - Kwale eye hospital, Mombasa
  - Kenyatta National Hospital, Nairobi
  - Lions SightFirst Hospital, Nairobi

IPD SHARING:
Plan to Share IPD: No